CLINICAL TRIAL: NCT00632125
Title: Post-authorization Safety Study to Prospectively Monitor the Incidence of Relevant Drug-related Adverse Events and EPO-related Lack of Efficacy Among CKD Subjects Receiving HX575 Recombinant Human Erythropoietin Alfa i.v.
Brief Title: Post-authorization Safety Study in CKD Subjects Receiving HX575 i.v.
Acronym: EPO-PASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-66-INJ-14
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Chronic Kidney Disease
Keywords: CKD subjects with or without dialysis treatment
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HX575 epoetin alfa i.v. (Experimental): This post-authorization safety study was designed as a multi-center, multinational, prospective, single-arm clinical study with a 6-month HX575 (recombinant human) erythropoietin alfa treatment period. It was planned to include approximately 1,500 patients.
  Interventions: Drug: HX575 recombinant human erythropoietin alfa

INTERVENTIONS:
Drug: HX575 recombinant human erythropoietin alfa — HX575 epoetin alfa i.v. will be administered according to the SmPC
  Other Names: HX575 epoetin alfa

SUMMARY:
Cumulative follow-up with HX575 epoetin alfa to prospectively monitor the incidence of relevant drug-related adverse events and EPO-related lack of efficacy among Chronic Kidney Disease (CKD) subjects receiving HX575 epoetin alfa i.v.

DETAILED DESCRIPTION:
This study was a multi-center, multinational, prospective, single-arm clinical study with a 6-month treatment period. The primary objective was to extend the safety database of patients with CKD who receive i.v. HX575 epoetin alfa treatment and to monitor the adverse event (AE) profile under post-approval conditions.

ELIGIBILITY:
Inclusion Criteria:

* CKD subjects with or without dialysis treatment
* Age over 18 years
* Subjects requiring i.v. ESA treatment
* Subjects likely to remain on i.v. ESA treatment for 6 months
* Provision of informed consent -

Exclusion Criteria:

* Systemic immunosuppressive medication or any other drugs known to adversely affect the hemoglobin level
* Known primary lack of efficacy (LOE), unexplained loss of effect to a recombinant erythropoietin product
* History of PRCA or aplastic anemia
* History of anti-erythropoietin antibodies
* Uncontrolled hypertension
* Pregnant woman or nursing mother
* Women of childbearing potential do not agree to maintain effective birth control during the study treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1695 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Roth, Dr, Study Chair — Hexal AG
Locations (114):
- Austria (5):
  - Dialysepraxis Dres. Huspek/Schmid, Bad Ischl
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Landeskrankenhaus Freistadt, Freistadt
  - LKH Rohrbach, Rohrbach
  - Universitätsklinik für Innere Medizin III, Vienna
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment Dr. Tota Venkova, Gabrovo
  - Multiprofile Hospital for Active Treatment Dr. Kiro Popov, Karlovo
  - Multiprofile Hospital for Active Treatment Pazardzhik, Pazardzhik
  - Multiprofile Hospital for Active Treatment Rousse, Rousse
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski, Sofia
  - Ministry of Interior-Central Clinical Base, Sofia
- CHG Hopital Yves le Foll, Saint-Brieuc, France
- Germany (40):
  - Fachpraxis für Nieren und Hochdruckerkrankungen, Andernach
  - KfH Kuratorium für Nierentranplantation und Dialyse e.V., Aschaffenburg
  - Gemeinschaftspraxis, Baunatal
  - Kuratorium ür Dialyse und Nierentransplantation e.V., Bayreuth
  - KfH Nierenzentrum, Berlin
  - Alwall Praxis für Nieren- und Hochdruckkrankheiten, Berlin
  - Dialysepraxis, Bremerhaven
  - Dialysepraxis Drs. Riedasch/Schreiber, Coesfeld
  - KfH Nierenzentrum, Cologne
  - Facharzt für Innere Medizin und Nephrologie, Dialyse Centrum, Darmstadt
  - KfH Kuratorium für Nierentranplantation und Dialyse e.V., Deggendorf
  - Dialysezentrum, Dinkelsbühl
  - Diabetes- und Dialysezentrum Merker, Vogt, Dormagen
  - KfH Nierenzentrum, Dortmund
  - Gemeinschaftspraxis Karlstraße, Düsseldorf
  - Kuratorium für Dialyse und Nierentransplantation e.V., Ehingen
  - Dialysezentrum Elsenfeld, Elsenfeld
  - Gemeinschaftspraxis Dr. Spitthöver, Dr. Knee, Dr. Gröschel, Essen
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V., Essen
  - Dialysezentrum, Freiburg im Breisgau
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Fürstenzell
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Gummersbach
  - Dialyse Hamburg Barmbek, Hamburg
  - Dialysepraxis Dr. Spengler, Helmstedt
  - Marienhospital Herne, Herne
  - Dialyse-Zentrum Elsterland, Herzberg
  - Praxis Dr. Menzer, Homberg (Efze)
  - Nephrologische Praxis, Höchstadt an der Aisch
  - Gemeinschaftspraxis, Kamp-Lintfort
  - Dialysepraxis, Lahr
  - Praxis für Innere Medizin und Nephrologie, Leverkusen
  - Nephrologisches Zentrum Emsland, Lingen
  - Dialysezentrum und Schwerpunktpraxis für Nieren- und Hochdruckerkrankungen, Mannheim
  - Gemeinschaftspraxis, Mayen
  - Nephrologisches Zentrum Mettmann, Mettmann
  - KfH Kuratorium für Nierentranplantation und Dialyse e.V., Oberschleißheim
  - Nierenzentrum Prenzlau, Prenzlau
  - Nephrologische Ambulanz/ Dialyse, Singen
  - KfH Kuratorium für Dialyse und Nierentransplantation e.V, Straubing
  - Nieren- und Diabeteszentrum Viersen-Nettetal, Viersen-Dülken
- Italy (22):
  - IRCCS INRCA Sede de Ancona, Ancona
  - Ospedali Riuniti di Anzio e Nettuno, Anzio
  - U.O.C. Nefrologia e Dialisi, C.G. Mazzoni, Ascoli Piceno
  - Ospedaliero Universitaria Policlinico S. Orsola Malpighi, Bologna
  - Azienda Ospdealiero "Istituti Ospitalieri", Cremona
  - Ospedale E. Profili di Fabriano, Fabriano
  - AO Universitaria Ospedali Riuniti, Foggia
  - Universitaria Degli Studi di Genova Clinica Nefrologica, Dialisi e Trapianto, Genova
  - Ospedale A. Manzoni, Lecco
  - Azienda Ospedaliera Carlo Poma di Mantova, Mantova
  - Azienda Ospedaliera Ospedale San Carlo Borromeo, Milan
  - Azienda Ospedaliera Ospedale Niguarda Ca Granda, Milan
  - AO Universitaria di Modena, Modena
  - Ospedale Maggiore di Modica, Modica
  - U.O. Nefrologia e Dialisi, P.O. Ospedale Casati, Centro Dialisi, Passirana Di Rho
  - Fondazione S. Maugeri, Pavia
  - Azienda Ospedaliera ospedale S. Salvatore, Pesaro
  - Ospedale A. Landolfi, Solofra
  - Azienda Ospedaliera CTO - Maria Adelaide, Torino
  - Ospedale San Giovanni Bosco, Torino
  - Ospedale di Trento / Santa Chiara, Trento
  - Ospedale dell'Angelo, Venezia Mestre
- North Macedonia (8):
  - PHO Clinical Hospital Dr. Trifun Panovski, Bitola
  - PHO Health organisation Goce Delcev, Delcevo
  - PHO General Hospital Kocani, Kočani
  - PHO General Hospital Borka Taleski, Prilep
  - PHO General Hospital Stip, Shtip
  - PHO Clinic of Nephrology, Skopje
  - Institute of Nephrology, Struga
  - PHO Medical Center Veles, Veles
- Poland (15):
  - Specjalistyczny Szpital Wojewodzki w Ciechanowie, Ciechanów
  - Wojewodzki Szpital Specjalistyczny im. Najswietszej maryi Panny, Częstochowa
  - Samodzielnym Publicznym Zakladzie Opieki Zdrowotnej Dzialdowo, Działdowo
  - Stacja Dializ w Garwolinie, Garwolin
  - Szpital Specjalistyczny Sw. W. Adalberta, Gdansk
  - Niepubliczny Zaklad Opieki Zdrowotnej AVITUM, Golub-Dobrzyń
  - B. Braun AVITUM Poland Sp., Legnica
  - SP Szpital Kliniczny im. Barlickiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin
  - Niepubliczny Zaklad Opieki Zdrowotnej, Pabianice
  - Radomski Szpital Specjalistyszny im. Dr Tytusa Chalubinskiego, Radom
  - Wojewodzki Szpital Specjalistyczny nr 3, Rybnik
  - Szpital Bielanski Blok F, Warsaw
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Szpital Powiatowy im. Lekarza Z. Koprowskiego, Warsaw
- Romania (5):
  - Spitalul Clinic Municipal, Arad
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Clinic de urgenta "Floreasca", Bucharest
  - Spitalul Universitar de Urgenta, Bucharest
  - SC Renamed Nefrodial SRL, Oradea
- Russia (4):
  - FGUZ Clinical hospital No. 83 of FMBA of Russia, Moscow
  - City Clinal Hospital # 34, Novosibirsk
  - MLPU "Clinical City Hospital # 1", Smolensk
  - GUZ "Yaroslavl regional clinical hospital", Yaroslavl
- Ukraine (8):
  - Oblasna klinichna likarnia imeni I.I.Mechnikova, Dnipropetrovsk
  - Oblasnyi tsentr urologii ta nefrologii, Kharkiv
  - Tsentralnyi miskyi klinichnyi hospital, Viddilennia gemodializu, Kyiv
  - Miska klinichna likarnia#3, Miskyi nefrologichnyi tsentr, Kyiv
  - Instytut nefrologii AMN Ukrainy viddil nefrologii ta dializu, Kyiv
  - Mykolaivska Oblasna Klinichna Likarnia, Viddilennia Gemodializu, Mykolayiv
  - Ternopilska Oblasna Klinichna Likarnia, Viddilennia Nefrologii ta Gemodializu, Ternopil
  - Oblasna klinikchna likarnia, tsentr transplantologii ta gemodializu, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Horl WH, Locatelli F, Haag-Weber M, Ode M, Roth K; Epo-PASS study group. Prospective multicenter study of HX575 (biosimilar epoetin-alpha) in patients with chronic kidney disease applying a target hemoglobin of 10--12 g/dl. Clin Nephrol. 2012 Jul;78(1):24-32. doi: 10.5414/cn107440. PMID 22732334

RESULTS

PARTICIPANT FLOW:
Groups:
- HX575: HX575 recombinant human erythropoietin alfa: HX575 epoetin alfa i.v. will be administered according to the summary of product characteristics (SmPC)
Period: Overall Study
Arm/Group | HX575
Started | 1695 (1,698 patients were enrolled but 3 patients did not receive any study medication.)
Completed | 1393
Not Completed | 302
Not completed — Death | 82
Not completed — Withdrawal by Subject | 44
Not completed — Adverse Event | 36
Not completed — Renal transplantation | 17
Not completed — Need for systemic immunosuppressive medi | 8
Not completed — Non-compliance | 8
Not completed — Development of uncontrolled hypertension | 5
Not completed — Moved to other dialysis unit, etc. | 102

BASELINE CHARACTERISTICS:
Groups:
- HX575: HX575 recombinant human erythropoietin alfa: HX575 epoetin alfa i.v. will be administered according to the SmPC
Arm/Group | HX575
Number analyzed (Participants) | 1695
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 737
  Male | 958
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 1671
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  Austria | 44
  Russian Federation | 29
  Romania | 103
  Macedonia, The Former Yugoslav Republic of | 143
  Ukraine | 204
  Poland | 220
  Italy | 205
  Bulgaria | 45
  France | 1
  Germany | 701

OUTCOME MEASURES:

1. Primary Outcome: Drug-related Adverse Events Consisting of Epoetin Alfa-induced Immunogenicity and Resulting Clinical Effects
Description: The incidence of relevant drug-related adverse events consisting of Epoetin alfa-induced immunogenicity and resulting blockade in erythroid maturation (e.g. pure red cell aplasia) and lack of efficacy
Time Frame: 6 months
Population: Safety population: The safety population consists of all patients that received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HX575: HX575 administered i.v. according to the SmPC
Arm/Group | HX575
Number analyzed (Participants) | 1695
percentage of participants
  Drug-related AEs | 7 [5.9 to 8.3]
  EPO-related lack of efficacy events | 0.18 [0.04 to 0.52]

ADVERSE EVENTS:
Arm/Group | HX575
All-Cause Mortality (participants affected / at risk) | 82/1695
Serious Adverse Events (participants affected / at risk) | 456/1695
Other Adverse Events (participants affected / at risk) | 1314/1695
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 (N=1695)
Pneumonia (Infections and infestations) | 34 (35)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 24 (28)
Atrial fibrillation (Cardiac disorders) | 13 (14)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 (11)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (11)
Pyrexia (General disorders) | 8 (8)
Cerebrovascular accident (Nervous system disorders) | 9 (9)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Arteriovenous fistula operation (Surgical and medical procedures) | 7 (8)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Haematuria (Renal and urinary disorders) | 2 (2)
Blood glucose fluctuation (Investigations) | 2 (2)
Cataract (Eye disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (5)
Amyloidosis (Immune system disorders) | 2 (2)
Bipolar I disorder (Psychiatric disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 2 (2)
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1)
Immobilisation prolonged (Social circumstances) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Sepsis (Infections and infestations) | 16 (16)
Bronchitis (Infections and infestations) | 9 (9)
Cellulitis (Infections and infestations) | 6 (6)
Gastroenteritis (Infections and infestations) | 5 (5)
Diverticulitis (Infections and infestations) | 4 (4)
Gangrene (Infections and infestations) | 4 (4)
Bronchopneumonia (Infections and infestations) | 3 (3)
Infection (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Urosepsis (Infections and infestations) | 3 (3)
Viral infection (Infections and infestations) | 3 (3)
Diabetic foot infection (Infections and infestations) | 2 (2)
Endocarditis (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 2 (2)
Osteomyelitis (Infections and infestations) | 2 (2)
Shunt infection (Infections and infestations) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 2 (2)
Abscess (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Candida sepsis (Infections and infestations) | 1 (1)
Cardiac valve abscess (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Catheter sepsis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Clostridium difficile sepsis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Diabetic gangrene (Infections and infestations) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1)
Infected cyst (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Pyothorax (Infections and infestations) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1)
Scrotal abscess (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 17 (17)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 11 (13)
Femoral neck fracture (Injury, poisoning and procedural complications) | 8 (8)
Shunt occlusion (Injury, poisoning and procedural complications) | 8 (8)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 6 (7)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 3 (4)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 3 (3)
Concussion (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2)
Shunt malfunction (Injury, poisoning and procedural complications) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Device breakage (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Pacemaker complication (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (2)
Cardiac failure (Cardiac disorders) | 11 (13)
Cardiac arrest (Cardiac disorders) | 10 (10)
Myocardial infarction (Cardiac disorders) | 10 (10)
Coronary artery disease (Cardiac disorders) | 6 (6)
Acute coronary syndrome (Cardiac disorders) | 5 (5)
Angina pectoris (Cardiac disorders) | 5 (5)
Acute myocardial infarction (Cardiac disorders) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 4 (4)
Aortic valve stenosis (Cardiac disorders) | 3 (3)
Tachyarrhythmia (Cardiac disorders) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 3 (3)
Atrioventricular block (Cardiac disorders) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Left ventricular failure (Cardiac disorders) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Aortic valve sclerosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 6 (7)
Vomiting (Gastrointestinal disorders) | 5 (5)
Gastritis (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 3 (3)
Faecaloma (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 3 (3)
Peritonitis (Gastrointestinal disorders) | 3 (3)
Subileus (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Gastric haemorrhage (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (10)
Hypotension (Vascular disorders) | 5 (5)
Extremity necrosis (Vascular disorders) | 4 (4)
Venous thrombosis (Vascular disorders) | 4 (4)
Circulatory collapse (Vascular disorders) | 3 (3)
Steal syndrome (Vascular disorders) | 3 (3)
Angiopathy (Vascular disorders) | 2 (3)
Arterial occlusive disease (Vascular disorders) | 2 (2)
Arteriosclerosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2)
Air embolism (Vascular disorders) | 1 (1)
Cardiovascular insufficiency (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Diabetic macroangiopathy (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Ischaemic limb pain (Vascular disorders) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm ruptured (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1)
Chest pain (General disorders) | 6 (6)
Sudden death (General disorders) | 6 (6)
Catheter related complication (General disorders) | 5 (6)
General physical health deterioration (General disorders) | 4 (4)
Multi-organ failure (General disorders) | 2 (2)
Sudden cardiac death (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1)
Catheter site pain (General disorders) | 1 (1)
Catheter thrombosis (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Cyst rupture (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Orthostatic intolerance (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 3 (3)
Aphasia (Nervous system disorders) | 2 (2)
Brain oedema (Nervous system disorders) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 2 (2)
Dementia (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 5 (5)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (3)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Catheter placement (Surgical and medical procedures) | 2 (2)
Leg amputation (Surgical and medical procedures) | 2 (2)
Parathyroidectomy (Surgical and medical procedures) | 2 (2)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1)
Carotid artery stent insertion (Surgical and medical procedures) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1)
Catheter removal (Surgical and medical procedures) | 1 (1)
Coronary angioplasty (Surgical and medical procedures) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1)
Foot amputation (Surgical and medical procedures) | 1 (1)
High frequency ablation (Surgical and medical procedures) | 1 (1)
Medical device implantation (Surgical and medical procedures) | 1 (1)
Nephrectomy (Surgical and medical procedures) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 2 (2)
Bladder diverticulum (Renal and urinary disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1)
Renal disorder (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Angiogram peripheral (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1)
Paracentesis abdomen (Investigations) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 2 (2)
Amaurosis (Eye disorders) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Ulcerative keratitis (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1)
Chronic hepatitis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Cryoglobulinaemia (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575 (N=1695)
Bronchitis (Infections and infestations) | 136 (163)
Nasopharyngitis (Infections and infestations) | 100 (111)
Diarrhoea (Gastrointestinal disorders) | 161 (208)
Nausea (Gastrointestinal disorders) | 105 (148)
Vomiting (Gastrointestinal disorders) | 102 (121)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 223 (429)
Procedural hypotension (Injury, poisoning and procedural complications) | 111 (194)
Hypertension (Vascular disorders) | 174 (342)
Hypotension (Vascular disorders) | 145 (298)
Headache (Nervous system disorders) | 181 (299)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.